CLINICAL TRIAL: NCT00616395
Title: Effects of Diet on Metabolism, Body Composition, Brain Function in Infants/Children
Brief Title: Study of Early Infant Diet on Growth and Development
Acronym: Beginnings
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 07130
Record Dates: First submitted 2007-12-31; First posted 2008-02-15 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: Infant Nutrition; Soy Phytochemicals; Infant Body Composition; Brain Function; Cognition and Development; Healthy Infants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, urine, and stool may be collected from some study participants.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no grouping: IDE used for outcome measurement not for an intervention.
  Interventions: Device: No intervention

INTERVENTIONS:
Device: No intervention

SUMMARY:
The purpose of this study is to characterize physical growth, body composition, dietary intake, neurobehavioral development, and brain function of infants and children fed mostly breast-milk, milk-based formula or soy-based formula during their first year of life. Children are followed from age 2 months to age 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Infants
* Birth weight = 6 to 9 lbs
* Mostly fed breast milk, milk-based formula, soy-based formula
* Mother over 18 years of age

Exclusion Criteria:

* Unhealthy pregnancy
* Illness during pregnancy or for the child that could interfere with the study parameters

Ages: 1 Month to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy infants
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2002-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2025-06 (Actual)

PRIMARY OUTCOMES:
Growth and development | yearly, 1-6 years

CONTACTS AND LOCATIONS:
Overall Officials: Aline Andres, Ph.D., Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Leandro da Cruz L, Fiecke C, Reed B, Martinez A, Keck A, Fuenmayor A, Sobik S, Rowell AC, Moore MB, Bimali M, Williams DK, Andres A. Soy Protein-based Infant Formula Feeding association with Adolescent Growth, Body Composition, Cardiometabolic health and Pubertal Development in Comparison with Cow's Milk-Based Infant Formula and Human Milk Feeding. J Nutr. 2026 Jan 22:101376. doi: 10.1016/j.tjnut.2026.101376. Online ahead of print. PMID 41580087
- [Derived] Chen JR, Samuel HA, Shlisky J, Sims CR, Lazarenko OP, Williams DK, Andres A, Badger TM. A longitudinal observational study of skeletal development between ages 3 mo and 6 y in children fed human milk, milk formula, or soy formula. Am J Clin Nutr. 2023 Jun;117(6):1211-1218. doi: 10.1016/j.ajcnut.2023.04.002. Epub 2023 Apr 5. PMID 37028556
- [Derived] Sobik S, Sims CR, McCorkle G, Bellando J, Sorensen ST, Badger TM, Casey PH, Williams DK, Andres A. Early infant feeding effect on growth and body composition during the first 6 years and neurodevelopment at age 72 months. Pediatr Res. 2021 Jul;90(1):140-147. doi: 10.1038/s41390-020-01157-z. Epub 2020 Sep 22. PMID 32961547
- [Derived] Brink LR, Mercer KE, Piccolo BD, Chintapalli SV, Elolimy A, Bowlin AK, Matazel KS, Pack L, Adams SH, Shankar K, Badger TM, Andres A, Yeruva L. Neonatal diet alters fecal microbiota and metabolome profiles at different ages in infants fed breast milk or formula. Am J Clin Nutr. 2020 Jun 1;111(6):1190-1202. doi: 10.1093/ajcn/nqaa076. PMID 32330237
- [Derived] Andres A, Moore MB, Linam LE, Casey PH, Cleves MA, Badger TM. Compared with feeding infants breast milk or cow-milk formula, soy formula feeding does not affect subsequent reproductive organ size at 5 years of age. J Nutr. 2015 May;145(5):871-5. doi: 10.3945/jn.114.206201. Epub 2015 Mar 11. PMID 25761499
- [Derived] Andres A, Casey PH, Cleves MA, Badger TM. Body fat and bone mineral content of infants fed breast milk, cow's milk formula, or soy formula during the first year of life. J Pediatr. 2013 Jul;163(1):49-54. doi: 10.1016/j.jpeds.2012.12.067. Epub 2013 Feb 1. PMID 23375908